CLINICAL TRIAL: NCT00356278
Title: A Cognitive Enhancer May Facilitate Behavioral Exposure Therapy for Veterans With PTSD
Brief Title: D-cycloserine and Virtual Reality Exposure to Treat Iraq War Veterans With PTSD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor in Psychiatry and Associate Vice Chair of Clinical Research, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00024846; DATR AD-TS (Other: Other); R01MH070880 (NIH)
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Stress Disorder, Post Traumatic
Keywords: D-Cycloserine; Virtual Reality; Exposure Therapy; Veterans; Cognitive Behavior Therapy; Translational Research
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cycloserine; Alprazolam; Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Participants will receive VRE therapy and D-cycloserine
  Interventions: Drug: D-Cycloserine; Behavioral: Virtual Reality Exposure Therapy
- B (Active Comparator): Participants will receive VRE therapy and alprazolam
  Interventions: Drug: Alprazolam; Behavioral: Virtual Reality Exposure Therapy
- C (Placebo Comparator): Participants will receive VRE therapy and placebo
  Interventions: Behavioral: Virtual Reality Exposure Therapy; Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine — D-Cycloserine doses will be 50 mg. There will be 5 pills total during study, each given 30 minutes prior to each VRE session.
  Arms: A
Drug: Alprazolam — Alprazolam doses will be 0.25 mg. There will be 5 pills total during study, each given 30 minutes prior to each VRE session.
  Other Names: Xanax
  Arms: B
Behavioral: Virtual Reality Exposure Therapy — VRE includes viewing scenes of virtual Iraq via a head mounted display. Other stimuli presented include sounds, smells and vibration. Each session will be 60 minutes with approximately 30 to 45 minutes of that wearing head mounted display.
Drug: Placebo — Placebo will be administered in the same manner as the active drugs.
  Arms: C

SUMMARY:
This study will determine whether a combination of virtual reality exposure therapy and D-cycloserine will reduce post-traumatic stress disorder symptoms in Iraq war veterans.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a type of anxiety disorder affecting people who have witnessed or experienced a traumatic event. Veterans of war are at an increased risk for developing PTSD because of their experiences with war and combat. Symptoms of PTSD often include flashbacks or nightmares, depression, anxiety or uneasiness, and feeling emotionally numb or distant toward others. Fortunately, PTSD can be treated, usually with some combination of anti-depressants, anti-anxiety medication, and therapy. Virtual reality exposure (VRE) therapy is a new type of treatment that helps people to overcome anxiety about trauma by facing situations with the use of virtual reality. D-cycloserine is a medication that has been found to enhance the effects of psychotherapy in recent studies. This study will determine the effectiveness of VRE therapy plus D-cycloserine at reducing PTSD symptoms in Iraq war veterans.

During this study, all participants will undergo one educational session and five VRE sessions. The first session will involve gathering information, learning common reactions to trauma, and participating in a breathing relaxation approach. The following five sessions will involve reviewing memories of Iraq and watching virtual Iraq sequences. Each participant will wear a head-mounted display during which they will view scenario settings such as cities, humvee convoys, and scenes related to combat. Participants will be randomly assigned to receive D-cycloserine, alprazolam (anti-anxiety drug), or placebo one half-hour before each VRE session.

Prior to the first treatment session, participants will undergo a startle reaction procedure. This will entail hearing sudden tones that last a fraction of a second, and viewing virtual reality scenes. Three small electrodes, attached to each participant's face, will measure the number of eye blinks during the procedure. At several times throughout the study, heart rate and skin conductance will also be measured with electrodes. Collection of saliva samples and measurement of blood pressure will also occur several times during this study. Before, during, and immediately after treatment, participants will complete questionnaires. Participants will be contacted 3, 6, and 12 months after treatment to assess symptoms and to schedule a time for an interview, additional questionnaires, and the virtual reality-based assessment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for PTSD due to Iraq military trauma
* Speaks English
* Healthy overall

Exclusion Criteria:

* History of mania, schizophrenia, or other psychoses
* Suicidal
* Current alcohol or drug dependence
* Medication free within 2 weeks of study entry for any medication that has been taken less than daily for the past month and medicine free within 4 weeks of study entry for any anxiolytic medication that has been taken daily for the last month or more
* Pregnant
* Special medical conditions, such as kidney insufficiency, chronic diseases, or history of significant head injury
* Stabilized on potentially data obscuring medication such as glucocorticoids

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2006-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O. Rothbaum, PhD, ABPP, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Rauch SAM, Koola C, Post L, Yasinski C, Norrholm SD, Black K, Rothbaum BO. In session extinction and outcome in Virtual Reality Exposure Therapy for PTSD. Behav Res Ther. 2018 Oct;109:1-9. doi: 10.1016/j.brat.2018.07.003. Epub 2018 Jul 20. PMID 30059794
- [Derived] Norrholm SD, Jovanovic T, Gerardi M, Breazeale KG, Price M, Davis M, Duncan E, Ressler KJ, Bradley B, Rizzo A, Tuerk PW, Rothbaum BO. Baseline psychophysiological and cortisol reactivity as a predictor of PTSD treatment outcome in virtual reality exposure therapy. Behav Res Ther. 2016 Jul;82:28-37. doi: 10.1016/j.brat.2016.05.002. Epub 2016 May 7. PMID 27183343
- [Derived] Rothbaum BO, Price M, Jovanovic T, Norrholm SD, Gerardi M, Dunlop B, Davis M, Bradley B, Duncan EJ, Rizzo A, Ressler KJ. A randomized, double-blind evaluation of D-cycloserine or alprazolam combined with virtual reality exposure therapy for posttraumatic stress disorder in Iraq and Afghanistan War veterans. Am J Psychiatry. 2014 Jun;171(6):640-8. doi: 10.1176/appi.ajp.2014.13121625. PMID 24743802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were self-referred or referred by professionals. Some patients were referred from both VA personnel and non-VA sources between January 2007-May 2013.
Groups:
- VRE Therapy and D-cycloserine: D-Cycloserine: D-Cycloserine doses will be 50 mg. There will be 5 pills total during study, each given 30 minutes prior to each VRE session.
  Virtual Reality Exposure Therapy: VRE includes viewing scenes of virtual Iraq via a head mounted display. Other stimuli presented include sounds, smells and vibration. Each session will be 60 minutes with approximately 30 to 45 minutes of that wearing head mounted display.
- VRE Therapy and Alprazolam: Alprazolam: Alprazolam doses will be 0.25 mg. There will be 5 pills total during study, each given 30 minutes prior to each VRE session.
  Virtual Reality Exposure Therapy: VRE includes viewing scenes of virtual Iraq via a head mounted display. Other stimuli presented include sounds, smells and vibration. Each session will be 60 minutes with approximately 30 to 45 minutes of that wearing head mounted display.
- VRE Therapy and Placebo: Virtual Reality Exposure Therapy: VRE includes viewing scenes of virtual Iraq via a head mounted display. Other stimuli presented include sounds, smells and vibration. Each session will be 60 minutes with approximately 30 to 45 minutes of that wearing head mounted display.
  Placebo: Placebo will be administered in the same manner as the active drugs.
Period: Overall Study
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Started | 53 | 50 | 53
Completed | 28 | 35 | 34
Not Completed | 25 | 15 | 19
Not completed — Withdrawal by Subject | 25 | 15 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo | Total
Number analyzed (Participants) | 53 | 50 | 53 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 50 | 53 | 156
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 49 | 49 | 50 | 148
Region of Enrollment [Number; unit: participants]
  United States | 53 | 50 | 53 | 156

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: Scores may range from 0 (no symptoms) to 136 (severe symptoms). The score is based on the first 17 CAPS items administered.
Time Frame: Baseline
Population: Intent to Treat Analyses using all available information with Full Information Maximum Likelihood Estimation (FIML)to handle missing data
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 85.3 [79.3 to 91.9] | 88 [82.3 to 93.6] | 82.6 [75.8 to 89.4]

2. Secondary Outcome: PTSD Symptom Scale Self-Report
Description: PTSD Symptom Scale - Self-Report Version (PSS-SR) is a 17-item self-reported questionnaire to assess symptoms of PTSD. Each of the 17 items describe PTSD symptoms which respondents rate in terms of their frequency or severity using a Likert-type scale ranging from 0 (not at all or only one time) to 3 (almost always or five or more times per week). Ratings on items are summed to create three subscales, including re-experiencing, avoidance, and arousal, as well as a total score (that ranges from 0 to 51). The total score higher than 13 indicates on likelihood of PTSD.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 32.9 [29.7 to 36.2] | 32.4 [26.0 to 38.9] | 32.4 [29.1 to 35.7]

3. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: Posttreatment, 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 65.9 [60.2 to 71.6] | 69.6 [63.8 to 75.4] | 63.8 [56.7 to 70.9]

4. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 60.3 [54.4 to 66.2] | 66.8 [59.6 to 74.0] | 51.5 [43.6 to 59.5]

5. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 56.0 [50.1 to 62.0] | 63.4 [55.4 to 71.4] | 46.9 [38.7 to 55.1]

6. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: as for outcome 1
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 48.0 [41.0 to 55.0] | 57.2 [50.6 to 63.8] | 48.4 [41.0 to 55.8]

7. Secondary Outcome: PTSD Symptom Scale Self-Report
Description: as for outcome 2
Time Frame: Posttreatment, 8 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 27.1 [24.3 to 29.9] | 25.6 [22.5 to 28.7] | 24.2 [20.2 to 28.1]

8. Secondary Outcome: PTSD Symptom Scale Self-Report
Description: as for outcome 2
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 25.2 [22.0 to 28.5] | 26.1 [22.6 to 29.4] | 21.4 [17.1 to 25.6]

9. Secondary Outcome: PTSD Symptom Scale Self-Report
Description: as for outcome 2
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 24.1 [20.5 to 27.6] | 26.3 [22.5 to 30.1] | 20.0 [15.9 to 24.0]

10. Secondary Outcome: PTSD Symptom Scale Self-Report
Description: as for outcome 2
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Number analyzed (Participants) | 53 | 50 | 53
units on a scale | 22.6 [19.1 to 26.1] | 24.2 [20.8 to 27.6] | 21.7 [17.9 to 25.4]

ADVERSE EVENTS:
Arm/Group | VRE Therapy and D-cycloserine | VRE Therapy and Alprazolam | VRE Therapy and Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50 | 0/53

LIMITATIONS AND CAVEATS:
The study had a high dropout rate. 31 participants dropped out before the first treatment session. Although disheartening, the dropout rate is similar to rates in other studies with veterans and active duty personnel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No